CLINICAL TRIAL: NCT04460196
Title: Healthcare Renunciation During the Confinement Period in Connection With the COVID-19 Epidemic in Adult Emergency Departments
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC20_0155
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-07

CONDITIONS: Emergency Medicine
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Each admitted patient will complete a questionnaire

SUMMARY:
Healthcare renunciation is defined as: "Individuals give up care when they do not seek services and health care professionals when they experience a disorder, experience a physical or mental disorder, or when they do not access all of the prescribed care." In 2008, 16.5% of the general French population reported having renounced care. The causes mentioned of the renunciation are mainly the financial difficulties, the deadlines of appointments considered too long, the geographical remoteness. In the department of Sarthe, the rate of cessation of care is estimated at 27.6% over the period from 2014 to 2017.

In the context of the COVID-19 epidemic, containment was applied in France counted from 17 March 2020. The widespread message was "save lives, stay at home". The Ministry of Solidarity and Health has provided health professionals with a circular to adapt the management of patients with chronic disease, requiring elective surgical care and pregnant women.

The decline in activity of general practitioners is estimated at 44% and that of other specialists at 71%. In Paris, visits to the emergency room fell by 45% for adults and 70% for children.

The main risk is the deterioration of the health status of some patients with the worsening of chronic diseases, the discovery of pathologies during episodes of decompensation and the absence of management of serious acute pathologies.

The study aims to assess the importance of giving up care during this period of COVID-19 and in comparison with a study conducted at the University Hospital of Angers and the hospital of Le Mans in 2017.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients consulting in the emergency department and agreeing to answer the questionnaire

Exclusion Criteria:

* Patient admitted in the emergency department in serious condition (life distress)
* Person unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person unable to give a non-opposition
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
rate of patients who gave up consulting in the emergency department | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Angers, Angers
  - CH Le Mans, Le Mans